CLINICAL TRIAL: NCT03713970
Title: Clinical Performance of Ceramic Laminate Veneers Made With Celtra Press and IPS e.Max Press Ceramic. Randomized Controlled Clinical Trial-one Year Evaluation
Brief Title: Clinical Performance of Ceramic Laminate Veneers Made With Celtra Duo Press and IPS e.Max Press Ceramic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, shafeq hashem saif aqlan, director, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-10-20
Record Dates: First submitted 2018-10-16; First posted 2018-10-22 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Fracture; Tooth Discoloration
Keywords: cetra duo press,e.max press,clinical performance
MeSH Terms: conditions — Fractures, Bone; Tooth Discoloration | interventions — IPS e.max Press

STUDY DESIGN:
Intervention Model Description: two groups withe different laminate veneers restorations(celtra duo press and IPS e.max press)
Who Masked: Participant, Care Provider, Investigator
Masking Description: After examining the participant for eligibility,each participant will be given a number start from one by Shafeq(the main researcher )i.e. each participant will be assigned by numbers and allocated to different groups using these numbers.(for example, the odd numbers to the intervention and the even numbers to the control group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celtra duo press (Experimental): Celtra duo press ingot 20g for three laminate veneers
  Interventions: Procedure: celtra duo press; Procedure: IPS e.max press
- IPS e.max press (Active Comparator): IPS e.max press ingot 20g for three laminate veneers
  Interventions: Procedure: celtra duo press; Procedure: IPS e.max press

INTERVENTIONS:
Procedure: celtra duo press — celtra duo press ingot
Procedure: IPS e.max press — IPS e.max press ingot

SUMMARY:
The aim of the present study is to assess the clinical performance (patient satisfaction, fracture, shade matching, Marginal adaptation and sensitivity) of laminate veneers made with celtra duo press ceramic and IPS e.max press ceramic with incisal wrap design.

DETAILED DESCRIPTION:
Ceramic materials are widely used for esthetic restorations because of their physical and optical properties that enhance patient satisfaction to dental restorations. several ceramic materials are currently available, including the lithium-reinforced glass ceramic like e.max press, which stands out for its excellent esthetic appearance and mechanical properties.also ZLS (zirconia-reinforced lithium silicate) are a function of its unique micro structure (500-700 nm in size, correspond exactly to the wavelength range of natural daylight). The presence of 10% zirconia in the glass phase in atomically dissolved form provides high strength and ensures safe and long-lasting restorations .The result is a large number of very fine-grained lithium silicate crystals, whose high glass content give the material its excellent light-optical and mechanical properties.

Translucency, opalescence, fluorescence and the chameleon effect all benefit, with high edge stability and excellent polishability being an added plus.3 Despite the recent introduction of improved ceramic materials, patient satisfaction with restoration contour,symmetry,margins and shade matching natural teeth with ceramic restorations is still one of the major challenges in clinical practice. The determination and interpretation of natural tooth color involve the selection and reproduction of ceramic shade and choice of restorative material. These factors have had a major influence on the final color of restorative treatments. Color-measuring instruments assist in shade analysis, thus minimizing the subjective variables of this process. Color readings allow improved determination of the restoration shade and better communication with the dental laboratory.4The influences of underlying substrate,8-9 luting agent,ceramic thickness and translucency, and restoration type14 on the color variation of ceramic restorations have been investigated in in vitro studies. Thus, the purpose of this study was to evaluate clinical performance of celtra duo press ceramic and IPS e.max press ceramic laminate veneers including patient satisfaction, fracture, shad matching, marginal adaptation and sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* All subjects were required to be
* at least 18 years old
* able to read and sign the informed consent document
* physically and psychologically able to tolerate conventional restorative procedures
* no active periodontal or pulpal diseases and teeth with good restorations
* teeth problems indicated for laminate veneer (e.g. discoloration, enamel fracture, chipping and mild malposition….)
* willing to return for follow-up examinations and evaluation
* Existing composite restorations of good quality, presenting no caries, ditching, or marginal staining were not removed prior to tooth preparation.
* normal bite (class I Kennedy classification)

Exclusion Criteria:

* Patients in the growth stage with partially erupted teeth
* fractured teeth of more than 50% enamel loss
* poor oral hygiene and motivation
* Pregnant women's
* endodontically treated teeth
* Psychiatric problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
color matching | 0ne year
  shad matching of both laminate veneers made with two materials compared to normal teeth will be evaluated using modified united state public health service criteria (USPHS) 0 Excellent colour match and shade between restoration and adjacent tooth, almost invisible.
  1 Slightly mismatching between the restoration and the adjacent tooth, which is in the normal range of tooth colour, translucence and/or shade.
  3 Obvious mismatch, beyond the normal range. 4 Gross mismatch/aesthetically displeasing colour, shade and/or translucence.

SECONDARY OUTCOMES:
fracture | one year
  fracture of dental laminate veneers made with two materials will be evaluated using modified united state public health service criteria (USPHS) 0 no fracture
  1. minor cracks line over the restoration
  2. minor chipping of the restoration (1/4)
  3. moderate chipping of the restoration (1/2)
  4. sever chipping of the restoration
  5. complete fracture
patient satisfaction | one year
  Primary objective to assess clinical performance (patient satisfaction) of laminate veneers made with celtra duo press ceramic and IPS e.max press ceramic with incisal wrap design using questionnaire.
  Questions
  Are you satisfied with new laminate? Are you satisfied with your laminate color? Have you noticed any color change in your crown till now? Do you feel that your laminate looks natural? Have you suffered from any kind of pain or problem during laminate use? Do you like your laminate alignment? Do you like your general appearance? Do you feel that the laminate is in harmony with the adjacent teeth? Have you experienced gingival or periodontal inflammation around the laminate after its insertion? Has the laminate stability affected through this year?
  the participant should be answer yes or no
Marginal adaptation | one year
  Marginal adaptation of both laminate veneers made with two materials will be evaluated using modified united state public health service criteria (USPHS) 0= smooth margin
  1. enamel exposed
  2. base or dentin exposed
  3. debonding from one end
  4. debonding from both ends
sensitivity | one year
  sensitivity of teeth that restored with laminate veneers made with two materials will be evaluated using modified united state public health service criteria (USPHS) 0 no sensitivity
  1. slight sensitivity
  2. moderate sensitivity
  3. sever sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- department of fixed prosthodontic-Cairo university, Cairo, Egypt

REFERENCES:
- [Result] Alhekeir DF, Al-Sarhan RA, Al Mashaan AF. Porcelain laminate veneers: Clinical survey for evaluation of failure. Saudi Dent J. 2014 Apr;26(2):63-7. doi: 10.1016/j.sdentj.2014.02.003. Epub 2014 Mar 26. PMID 25408598
- [Result] Chu SJ, Trushkowsky RD, Paravina RD. Dental color matching instruments and systems. Review of clinical and research aspects. J Dent. 2010;38 Suppl 2:e2-16. doi: 10.1016/j.jdent.2010.07.001. Epub 2010 Aug 1. PMID 20621154
- [Result] Stevenson B, Ibbetson R. The effect of the substructure on the colour of samples/restorations veneered with ceramic: a literature review. J Dent. 2010 May;38(5):361-8. doi: 10.1016/j.jdent.2010.01.009. Epub 2010 Feb 1. PMID 20122985